CLINICAL TRIAL: NCT02992717
Title: Validation of the 3D-CAM in the Recovery Room to Detect Postoperative Delirium Compared to Nu-DESC, CAM and DSM-5 Criteria
Brief Title: Validation of the 3D-CAM to Detect Postoperative Delirium
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charité - University Medicine Berlin, Charite University, Berlin, Germany
Other Study IDs: 3D_CAM
Record Dates: First submitted 2016-12-08; First posted 2016-12-14 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing elective general anaesthesia: Male and female adult patients undergoing elective general anaesthesia.

SUMMARY:
The 3D-CAM is a new 3-minute diagnostic assessment for Confusion Assessment Method-defined Delirium. The primary objective of this study is to translate the 3D-CAM into the German language, as well as to validate its use to detect postoperative delirium in the recovery room. The validation will be based on comparisons to the Nu-DESC (Nursing Delirium Screening Scale), CAM (Confusion Assessment Method), and DSM-5 criteria (Diagnostic and Statistical Manual of Mental Disorders).

DETAILED DESCRIPTION:
Approximately 200 patients will be enrolled in the study. They will followed up until the third postoperative day.

Calculation and analysis of demographic and perioperative influencing factors on postoperative delirium according to routine parameters (age, sex, body height, body weight, diagnosis, physical status according to the American Society of Anaesthesiologists (ASA PS), duration of surgery, Physiological and Operative Severity Score (POSSUM), type of anesthesia, medication against pain and delirium) will be performed.

ELIGIBILITY:
Inclusion criteria:

* Male and female patients with age ≥ 18 years
* Admission to recovery room (RR) or post anaesthesia care unit (PACU) following elective general anaesthesia and scheduled
* Inpatient treatment not less than 24 hours.

Exclusion criteria:

* Patients with psychiatric diseases and mental retardation
* Analphabetism
* Anacusis or Hypoacusis with hearing aid device,
* Amaurosis
* Lacking willingness to save and hand out data within the study
* Accommodation in an institution due to an official or judicial order
* Patients with unability speaking German or English language
* Participation in other clinical studies during the study period
* Coworker in the study site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female adult patients undergoing elective general anaesthesia.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the delirium screening/diagnosing tool "3D Confusion Assessment Method (3D-CAM) | Up to three days
  Sensitivity of the delirium screening/diagnosing tool "3D Confusion Assessment Method (3D-CAM)" to detect postoperative delirium (POD) in the recovery room - Used reference standard: DSM-5 criteria
Specificity of the delirium screening/diagnosing tool "3D Confusion Assessment Method (3D-CAM) | Up to three days
  Specificity of the delirium screening/diagnosing tool "3D Confusion Assessment Method (3D-CAM) to detect postoperative delirium (POD) in the recovery room - Used reference standard: DSM-5 criteria

SECONDARY OUTCOMES:
Test Quality Level | Up to three days
  Comparison of test Quality level between 3D-CAM, Nu-DESC and CAM to detect POD in the recovery room.
Duration of postoperative delirium | Up to three days
Duration of stay in recovery room | Up to three days
Duration of performance of the delirium testings | Up to three days
Pain level | Participants will be followed up until the third postoperative day
Postoperative complications | Up to three days
  Postoperative complications according to Clavien-Dindo classification
Duration of hospital stay | Participants will be followed for the duration of hospital stay an expected average of 3 weeks
In-house mortality | Participants will be followed for the duration of hospital stay an expected average of 3 weeks
Follow-up care | Participants will be followed for the duration of hospital stay an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Charité Mitte and Campus Virchow - Klinikum, Charite University, Berlin, Germany, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olbert M, Eckert S, Morgeli R, Kruppa J, Spies CD. Validation of 3-minute diagnostic interview for CAM-defined Delirium to detect postoperative delirium in the recovery room: A prospective diagnostic study. Eur J Anaesthesiol. 2019 Sep;36(9):683-687. doi: 10.1097/EJA.0000000000001048. PMID 31306183